CLINICAL TRIAL: NCT06522152
Title: Evaluation of Clinical-functional and Radiographic Outcomes in Patients Who Underwent Meniscal Allograft Transplantation (MAT) at 10 Years.
Acronym: MAT 10 Y
Status: Recruiting | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Principal Investigator, Stefano Zaffagnini, Full Professor Medicine and Surgery, University of Bologna, Istituto Ortopedico Rizzoli
Other Study IDs: MAT 10 Y
Record Dates: First submitted 2024-07-22; First posted 2024-07-26 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Meniscus Disorder; Arthritis Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Menisci are crescent-shaped cartilage structures that are fundamentally important for the biomechanics and physiology of the knee joint. They play a primary role in load transmission, assist the ligaments in ensuring knee stability, and thus protect against the onset of knee osteoarthritis. Meniscal injuries are the most frequently encountered joint pathology and can cause pain, mechanical blocks, and recurrent effusions. The treatment of these injuries has progressively evolved from meniscectomy (removal of damaged meniscal tissue) to the use of meniscal sutures (where possible) to allow the preservation of the greatest amount of meniscus: numerous studies have shown a correlation between the amount of meniscus removed and the future onset of osteoarthritis (Hutchinson AJSM 2014, Harston KSSTA 2012).

However, in some cases, especially in the presence of complex and/or chronic lesions, meniscectomy remains the only viable surgical solution even today. Over time, months or years later, a subgroup of patients experiences symptoms such as pain, joint swelling, and mechanical overload of the compartment subjected to meniscectomy, a condition known as "post-meniscectomy syndrome." Some of these patients will subsequently develop knee osteoarthritis, requiring invasive interventions such as partial or total knee replacement.

Meniscal allograft transplantation (MAT) represents a valid therapeutic option for post-meniscectomy syndrome. This procedure aims to restore joint functionality and stability through the transplantation of a meniscus from a cadaver donor. MAT has been widely adopted in clinical practice, showing success in reducing pain and improving joint functionality.

Current studies suggest that meniscal transplantation can offer significant protection against osteoarthritis, but the duration of this preventive effect is not yet fully understood. Furthermore, there are no studies that can demonstrate the state of osteoarthritis with radiographic controls pre- and post-treatment at a follow-up of over 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 65 at the time of surgery
* Both male and female
* Patients who underwent meniscal transplantation at the Rizzoli Orthopedic Institute at least 10 years ago

Exclusion Criteria:

* Patients who do not give consent to be included in the study
* Patients who are no longer reachable
* Presence of infection or hematologic, rheumatic, or coagulation disorders at the time of evaluation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 397 patients will be considered, recruited from all individuals who underwent meniscal transplantation at the Rizzoli Orthopedic Institute between June 2004 and October 2020, and who were previously recruited for the MAT study.
Sampling Method: Non-Probability Sample
Enrollment: 397 (Estimated)
Dates: Start 2024-10-24 (Actual); Primary Completion 2030-07 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
Lysholm Knee Score | 10 years
  It is a validated measurement scale that assesses knee functionality through 8 items, which allow for determining the condition of the knee in response to the functional demands of daily life activities. This evaluation form is used to assess the outcomes of surgery on patients operated on for ligamentous or meniscal knee injuries. The final score is obtained by summing the various scores obtained in the different items, ranging from 0 to 100. The scores are divided into subgroups: Excellent (95-100); Good (84-94); Fair (65-83); Poor (<64).
Kellgren-Lawrence scale | 10 years
  Clinical and imaging material in the patient's possession will be collected to evaluate the potential development of osteoarthritis. If the patient does not have radiological documentation performed according to the study protocol within the last 12 months, a weight-bearing knee X-ray in two projections will be performed to assess the degree of osteoarthritis according to the Kellgren-Lawrence scale.

SECONDARY OUTCOMES:
VAS | 10 years
  It is a 10-point quantitative unidimensional numerical scale for pain assessment. The scale requires the patient to select the number that best describes the intensity of their pain, from 0 to 10, at that precise moment. 0 means no pain, and 10 indicates the worst possible pain.
Tegner Score | 10 years
  It allows estimating the level of motor activity of a subject with a score between 0 and 10, where 0 represents 'inability' and 10 represents 'participation in competitive sports, such as national or international level soccer.' This score is the most commonly used to define the level of motor activity in patients with knee disorders. In the study, the Tegner Score will be completed directly by the investigator through an interview with the patient.
KOOS score | 10 years
  The Knee Injury and Osteoarthritis Outcome Score (KOOS) is a questionnaire aimed at assessing symptoms related to the knee joint in individuals with joint injuries or primary osteoarthritis. It evaluates knee functionality across 5 aspects: symptoms, pain, Activities of Daily Living (ADL), sports, and Quality of Life (QOL). The final score is obtained by summing the various scores from the different items and ranges from 0 to 100.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Istituto Ortopedico Rizzoli, Bologna, Italy